CLINICAL TRIAL: NCT03396653
Title: Peer Support for Weight Loss Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Stanford University (Other); The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Tricia Leahey, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H17-099; 1R01DK111232-01A1 (NIH)
Record Dates: First submitted 2017-12-29; First posted 2018-01-11 (Actual); Results first posted 2024-05-02 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Obesity
Keywords: weight loss; weight maintenance; weight control; peer support; patient-provided care
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-Delivered Weight Maintenance (Active Comparator): Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive an 18-month patient-delivered behavioral weight maintenance intervention. Specifically, group sessions will be delivered by a mentor (i.e., successful weight loser) and weekly coaching will be delivered by a peer (other member of their weight maintenance group).
  Interventions: Behavioral: Peer-delivered Weight Maintenance
- Professionally-Delivered Weight Maintenance (Active Comparator): Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive an 18-month reduced intensity behavioral weight maintenance intervention, delivered by a professional. The intervention will consist of 24 group sessions.
  Interventions: Behavioral: Professionally-Delivered Weight Maintenance

INTERVENTIONS:
Behavioral: Peer-delivered Weight Maintenance — Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive an 18-month patient-delivered behavioral weight maintenance intervention. Specifically, group sessions will be delivered by a mentor (i.e., successful weight loser) and weekly coaching will be delivered by a peer (other member of their weight maintenance group).
  Arms: Peer-Delivered Weight Maintenance
Behavioral: Professionally-Delivered Weight Maintenance — Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive an 18-month reduced intensity behavioral weight maintenance intervention, delivered by a professional. The intervention will consist of 24 group sessions.
  Arms: Professionally-Delivered Weight Maintenance

SUMMARY:
The primary aim of this study is to test the efficacy of patient-provided treatment for weight-loss maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75
* Body Mass Index between 25-50
* English Speaking

Exclusion Criteria:

* Report being unable to walk 2 blocks without stopping
* Are currently participating in weight loss treatment, have a history of bariatric surgery, or lost ≥5% in the past 6-months
* Are pregnant or plan to become pregnant within 1 year
* Report a heart condition, chest pain during periods of rest or activity, or loss of consciousness on the Physical Activity Readiness Questionnaire
* Report a medical condition that could jeopardize their safety in a weight control program with diet and exercise guidelines
* Report conditions that, in the judgment of the PI, would render them unlikely to follow the protocol (e.g., relocation, dementia, unable to read and write in English)
* Have no Internet access.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 849 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UConn's Weight Management Research Group, Hartford, Connecticut
  - Institute for Collaboration on Health, Intervention and Policy, Storrs, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leahey TM, Gorin AA, Huedo-Medina TB, Denmat Z, Field C, Gilder C, Wyckoff EP, O'Connor K, Hahn K, Jenkins K, Unick JL, Hand G, McManus-Shipp K, Calcaterra J, Falk G. Patient-Delivered Continuous Care for Weight Loss Maintenance: A Randomized Clinical Trial. JAMA Intern Med. 2025 Jul 1;185(7):767-776. doi: 10.1001/jamainternmed.2025.1345. PMID 40423949

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following enrollment, participants began Phase I, a 16-week weight loss program aiming to induce clinically significant weight loss (5% of starting body weight). After Phase I, eligibility to continue to Phase II (weight maintenance) was evaluated. Those who lost at least 5% of their body weight remained eligible. Given that Phase II was the primary focus of the study, primary outcome data were analyzed only from randomized, Phase II participants (eligible subset of Phase I participants).
Groups:
- Phase I: Weight Loss Phase and Phase II (RCT): Peer-Delivered Weight Maintenance: Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive an 18-month patient-delivered behavioral weight maintenance intervention. Specifically, group sessions will be delivered by a mentor (i.e., successful weight loser) and weekly coaching will be delivered by a peer (other member of their weight maintenance group).
  Peer-delivered Weight Maintenance: Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive an 18-month patient-delivered behavioral weight maintenance intervention. Specifically, group sessions will be delivered by a mentor (i.e., successful weight loser) and weekly coaching will be delivered by a peer (other member of their weight maintenance group).
- Phase I: Weight Loss Phase and Phase II (RCT): Professionally-Delivered Weight Maintenance: Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive an 18-month reduced intensity behavioral weight maintenance intervention, delivered by a professional. The intervention will consist of 24 group sessions.
  Professionally-Delivered Weight Maintenance: Contingent upon participants losing 5% of body weight or more in Phase I (weight loss) of this trial, participants will receive an 18-month reduced intensity behavioral weight maintenance intervention, delivered by a professional. The intervention will consist of 24 group sessions.
- Phase I Only (Weight Loss Phase): 16 Weeks: This group consists of the participants who enrolled in Phase I (Weight Loss Phase) but were not randomized to Phase I because they dropped out or were not eligible for Phase II (Weight Maintenance Phase).
Period: Phase I (Weight Loss): 16 Weeks
Arm/Group | Phase I: Weight Loss Phase and Phase II (RCT): Peer-Delivered Weight Maintenance | Phase I: Weight Loss Phase and Phase II (RCT): Professionally-Delivered Weight Maintenance | Phase I Only (Weight Loss Phase): 16 Weeks
Started | 153 | 134 | 562
Completed | 153 (For this Phase, completion would include 1) participation in the entire 16-week program 2) completion of the post-Phase I assessment and 3) confirmed eligible for Phase II. All participants in this arm were eligible and randomized into the Phase II Weight Maintenance RCT.) | 134 (For this Phase, completion would include 1) participation in the entire 16-week program 2) completion of the post-Phase I assessment and 3) confirmed eligible for Phase II. All participants in this arm were eligible and randomized into the Phase II Weight Maintenance RCT.) | 0 (For this Phase, completion would include 1) participation in the entire 16-week program 2) completion of the post-Phase I assessment and 3) confirmed eligible for Phase II. Because participants in this group did not meet all 3 of these requirements and were not randomized, all are considered incomplete.)
Not Completed | 0 | 0 | 562
Period: Phase II (Weight Maintenance): 18 Months
Arm/Group | Phase I: Weight Loss Phase and Phase II (RCT): Peer-Delivered Weight Maintenance | Phase I: Weight Loss Phase and Phase II (RCT): Professionally-Delivered Weight Maintenance | Phase I Only (Weight Loss Phase): 16 Weeks
Started | 153 | 134 | 0 (0)
6 Month Assessment | 145 | 131 | 0 (Participants in this group were not eligible for Phase II; therefore, these milestones are not applicable.)
12 Month Assessment | 139 | 122 | 0 (Participants in this group were not eligible for Phase II; therefore, these milestones are not applicable.)
Completed | 144 | 123 | 0 (Participants in this group were not eligible for Phase II; therefore, these milestones are not applicable.)
Not Completed | 9 | 11 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Weight Loss Phase and Phase II (RCT): Peer-Delivered Weight Maintenance | Phase I: Weight Loss Phase and Phase II (RCT): Professionally-Delivered Weight Maintenance | Phase I Only (Weight Loss Phase): 16 Weeks | Total
Number analyzed (Participants) | 153 | 134 | 562 | 849
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.6 (11.7) | 54.8 (11.7) | 48.9 (12.2) | 50.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 111 | 464 | 704
  Male | 24 | 23 | 98 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 18 | 94 | 125
  Not Hispanic or Latino | 140 | 116 | 434 | 690
  Unknown or Not Reported | 0 | 0 | 34 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 3
  Asian | 6 | 5 | 15 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 15 | 19 | 87 | 121
  White | 125 | 101 | 395 | 621
  More than one race | 7 | 5 | 16 | 28
  Unknown or Not Reported | 0 | 2 | 47 | 49
Region of Enrollment [Number; unit: participants]
  United States | 153 | 134 | 562 | 849
Weight (kg) [Mean (Standard Deviation); unit: kilograms] — Population: This study specific measure was first collected at Phase II baseline and data were analyzed only from randomized Phase II participants.
  kilograms
    number analyzed (Participants) | 153 | 134 | 0 | 287
    (all) | 82.9 (15.3) | 85.4 (17.4) |  | 84.0 (16.3)
Blood pressure (mmHg) [Mean (Standard Deviation); unit: mm Hg] — Population: This study specific measure was first collected at Phase II baseline and data were analyzed only from randomized Phase II participants.
  mm Hg
    Systolic Blood Pressure: number analyzed (Participants) | 153 | 134 | 0 | 287
    Systolic Blood Pressure | 118.6 (15.6) | 118.4 (13.2) |  | 118.5 (14.5)
    Diastolic Blood Pressure: number analyzed (Participants) | 153 | 134 | 0 | 287
    Diastolic Blood Pressure | 76.4 (8.3) | 76.8 (9.3) |  | 76.6 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Weight Change (kg)
Description: Weight change (measured on a digital scale to the nearest 0.1-kilogram) from Phase II Baseline (post-Phase I) to the end of the Phase II maintenance program (18 months).
Time Frame: Baseline to 18-months
Population: The number of participants analyzed in this outcome measure reflects the number that completed this measure at the 18 month assessment (primary outcome assessment). All missing participant data indicates that the participant did not complete this assessment procedure.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Peer-Delivered Weight Maintenance | Professionally-Delivered Weight Maintenance
Number analyzed (Participants) | 144 | 124
kilograms | 1.2 (7.0) | 2.5 (6.0)

2. Secondary Outcome: Blood Pressure (mmHg)
Description: Blood pressure (mmHg) from Phase II Baseline (post-Phase I) to the end of the Phase II maintenance program (18 months).
Time Frame: Baseline to 18-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Peer-Delivered Weight Maintenance | Professionally-Delivered Weight Maintenance
Number analyzed (Participants) | 141 | 122
mmHg
  Systolic Blood Pressure | 2.5 (13.4) | 4.0 (14.2)
  Diastolic Blood Pressure | 3.3 (8.2) | 4.6 (9.4)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for all participants enrolled in Phase I (including participants randomized to Phase II) from from the start of the program to the post-Phase I assessment (a total of 16 weeks). For participants randomized to Phase II, Adverse events data were additionally collected at the Phase II baseline, 6-month, 12-month, 18-month assessments, as well as the no-treatment follow up assessment at 24 months.
Arm/Group | Phase I: Weight Loss Phase and Phase II (RCT): Peer-Delivered Weight Maintenance | Phase I: Weight Loss Phase and Phase II (RCT): Professionally-Delivered Weight Maintenance | Phase I Only (Weight Loss Phase): 16 Weeks
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/134 | 0/562
Serious Adverse Events (participants affected / at risk) | 36/153 | 22/134 | 0/562
Other Adverse Events (participants affected / at risk) | 103/153 | 89/134 | 18/562
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Weight Loss Phase and Phase II (RCT): Peer-Delivered Weight Maintenance (N=153) | Phase I: Weight Loss Phase and Phase II (RCT): Professionally-Delivered Weight Maintenance (N=134) | Phase I Only (Weight Loss Phase): 16 Weeks (N=562)
Heart Trouble (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Muscle or bone injury (e.g., broken bone, torn ligament, sprain) (Injury, poisoning and procedural complications) | 7 (8) | 8 (8) | 0 (0)
Other (General disorders) | 19 (19) | 13 (13) | 0 (0)
Stroke, ministroke (TIA), or other neurological problems (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0)
Gall bladder attack or surgery (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
New diagnosis, started treatment, or hospitalized for depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma attack: leading to hospitalization or visit to ER / urgent care (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Fainting (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Weight Loss Phase and Phase II (RCT): Peer-Delivered Weight Maintenance (N=153) | Phase I: Weight Loss Phase and Phase II (RCT): Professionally-Delivered Weight Maintenance (N=134) | Phase I Only (Weight Loss Phase): 16 Weeks (N=562)
Heart Trouble (Cardiac disorders) | 10 (13) | 10 (13) | 1 (1)
Fainting (Nervous system disorders) | 9 (11) | 3 (3) | 0 (0)
Stroke, ministroke (TIA), or other neurological problems (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Muscle or bone injury (e.g., broken bone, torn ligament, sprain) (Injury, poisoning and procedural complications) | 39 (55) | 42 (65) | 9 (10)
New diagnosis or hospitalization for diabetes (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
New diagnosis, started treatment, or hospitalized for depression (Psychiatric disorders) | 3 (3) | 2 (2) | 1 (1)
Eating disorder (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1)
New diagnosis, started treatment or hospitalized for any other mental health problem (Psychiatric disorders) | 2 (2) | 3 (3) | 0 (0)
Asthma attack: leading to hospitalization or visit to ER / urgent care (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (2) | 0 (0) | 0 (0)
Weight loss medication (including herbal remedies) (Surgical and medical procedures) | 4 (4) | 3 (3) | 0 (0)
Motor vehicle accident (Injury, poisoning and procedural complications) | 11 (11) | 8 (8) | 1 (1)
Other (General disorders) | 75 (105) | 68 (104) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT03396653/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT03396653/ICF_001.pdf